CLINICAL TRIAL: NCT03725683
Title: A Prospective, Multicenter Study On the Effects of Progressive and Matched Caliber Balloon Predilation of Popliteal Artery On Treatment Strategy and Prognosis
Brief Title: Multi-center Study On the Treatment and Prognosis of Arteriosclerosis Obliterans With Different Caliber Balloon
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jun-min Bao (Network)
Responsible Party: Sponsor-Investigator, Jun-min Bao, chairman of the expert committee of lower limb artery disease, Chinese Medical Association
Organization: Chinese Medical Association (Network)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JUn-min Bao
Record Dates: First submitted 2018-10-22; First posted 2018-10-31 (Actual); Last update posted 2019-10-09 (Actual); Status verified 2019-10

CONDITIONS: Arteriosclerosis; Extremities
MeSH Terms: conditions — Arteriosclerosis

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Incrementing groups (Experimental): Each of the Increased caliber balloon capsules was predilated one by one, and the order of the increased balloon capsules was as follows: Balloon 2 diameter = target lesion reference vessel diameter minus 1; Balloon 3 diameter = target lesion reference vessel diameter;
  Interventions: Device: Increased caliber balloon
- matching groups (Experimental): Pre-dilatation of the matched caliber balloon, whose diameter = the target lesion's diameter as a reference vessel, was applied.
  Interventions: Device: matched caliber balloon

INTERVENTIONS:
Device: Increased caliber balloon — Imaging of target lesions was performed before surgery to evaluate the characteristics of target lesions.
  Postoperative to discharge Laboratory examination: blood routine, renal function, biochemical, coagulation functionTo determine and record the ABI(ankle-brachial pressure index);Records Rutherford classification; record the application of anticoagulant and antiplatelet agents; Records of adverse events.
  Arms: Incrementing groups
Device: matched caliber balloon — Imaging of target lesions was performed before surgery to evaluate the characteristics of target lesions.
  Postoperative to discharge Laboratory examination: blood routine, renal function, biochemical, coagulation functionTo determine and record the ABI index;Records Rutherford classification; record the application of anticoagulant and antiplatelet agents; Records of adverse events.
  Arms: matching groups

SUMMARY:
In the endoscopic treatment of superficial femoral artery and/or proximal popliteal artery in patients with lower extremity arteriosclerosis occlusion, the intercalation caused by the predilation of increasing caliber balloon and matching caliber balloon was compared, and then the impact of the two predilation methods on the intraoperative treatment strategy and short and medium-term prognosis was analyzed. The study was designed as a prospective, multi-center, single-blind, randomized, controlled study. It is planned to set up 5-10 research centers with 340 subjects, and the single center will be less than or equal to 100 subjects, in the form of competition from each research center.

ELIGIBILITY:
Inclusion Criteria:

1. Target lesions from superficial femoral artery to popliteal artery P1 segment; Proximal anatomical markers of target lesions:

   1. 1cm below the fork of the common femoral artery;
   2. Distal anatomical sign of target lesions: upper border of patella;
2. Target lesions may be single, combined, or tandem primary lesions of stenosis and/or occlusion, and meet one of the following criteria:

   1. In contrast, The stenosis rate was greater than or equal to 70% and less than 100%, and the total length of the lesions was greater than or equal to 40mm and less than or equal to 200mm.
   2. The total length of the lesion is less than 100mm.
   3. The total length of the lesion is less than or equal to 200mm, and the length of the occlusion segment is less than or equal to 100mm.

   Note: the distance between the lesions is no more than 30mm, and the distance between the lesions is > 30mm. Patients with multiple target lesions judged as 2 or more independent lesions met the inclusion criteria.
3. The diameter of the reference vessels of target lesions shall be 4mm or more and 7mm or less.
4. If the subject has ipsilateral iliac or lower knee lesions to be treated, the above lesions shall be successfully treated with target lesions, and the following criteria shall be met:

   1. Residual stricture of the common iliac lesion < 30%;
   2. An upper knee has at least one or more free outflow tract, i.e., residual stenosis < 50%;
   3. No embolism, rupture or other serious adverse events occurred during the operation.
5. The pregnancy test results of fertile female subjects must be negative and there is no pregnancy plan during the study period;
6. The patient or client signs the patient's informed consent;
7. Understand and accept the duration of this study, and be able to cooperate with follow-up and evaluation;
8. Subject's life expectancy is greater than or equal to 12 months after evaluation by the investigator.

Exclusion Criteria:

1. The investigator believes that the subject has the possibility of non-compliance with the follow-up plan;
2. Patients with cerebral apoplexy or st-segment elevation myocardial infarction in the last 3 months;
3. Combined with the following diseases

   1. Patients diagnosed with thrombotic occlusive vasculitis;
   2. combined with abdominal aortic aneurysm/thoraco-abdominal aortic aneurysm (with mural thrombus inside the aneurysm cavity);
   3. coagulation defect;
   4. high coagulation status;
4. blood index

   1. Serum creatinine > 170umol;
   2. White blood cell count < 3.0 x 109/L or > 14.0 x 109/L;
   3. Patients with platelet count < 80 x 109/L or > 500 x 109/L;
5. Patients who are known to be allergic to anticoagulant, antiplatelet, contrast agent and other drugs; Examples: heparin, clopidogrel, iodixanol, etc.
6. Target lesions are non-primary lesions of restenosis and anastomotic stenosis within the stent;
7. Acute or subacute thrombosis of target lesions;
8. There are aneurysms in the vicinity of target lesions, and the proximity refers to no more than 20mm.
9. The patient is a lactating woman or a pregnant woman.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2019-11-01 (Estimated); Primary Completion 2020-11-01 (Estimated); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
success rate of balloon repair | during the surgery
  During the surgery:successful conduction, accurate positioning and release, and no narrowing or blocking of the balloon. Immediately after the balloon release, angiography shows balloon patency, successful expansion of stenosis, and arteriorrhexis or dissection rupture.

SECONDARY OUTCOMES:
Balloon related adverse event rate | 7 days after operation
  Renal insufficiency due to surgery; Changes in coagulation function; Degree of arterial stenosis and Degree of limb ischemia；
  Other adverse events

OTHER OUTCOMES:
30days±7days related adverse event rate | 30days±7days
  Changes in coagulation function; Degree of arterial stenosis and Degree of limb ischemia； Other adverse events
6months±30days related adverse event rate | 6months±30days
  Changes in coagulation function; Degree of arterial stenosis and Degree of limb ischemia； Other adverse events
12months±30days related adverse event rate | 12months±30days
  Changes in coagulation function; Degree of arterial stenosis and Degree of limb ischemia； Other adverse events

CONTACTS AND LOCATIONS:
Locations (11):
- China (11):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Xuanwu Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Gulou Hospital, Nanjing, Jiangsu
  - Nanjing first hospital, Nanjing, Jiangsu
  - Shanghai Ninth People's Hospital, Shanghai, Shanghai Municipality
  - Shanghai Renji Hospital, Shanghai, Shanghai Municipality
  - Shanghai Zhongshan Hospital, Shanghai, Shanghai Municipality
  - Shanxi da Hospital, Taiyuan, Shanxi
  - The Affiliated Hospital of Southwest Medical University, Luzhou, Sichuan
  - People's Hospital of XinJiang Uygur Autonomous Region, Ürümqi, Xinjiang

IPD SHARING:
Plan to Share IPD: No